CLINICAL TRIAL: NCT05141149
Title: A First in Human, Phase 1/2a, Multicentre, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of PBP1510 in Patients With Advanced/Metastatic Pancreatic Cancer
Brief Title: First in Human Phase1/2a Clinical Trial of Anti-PAUF Monoclonal Antibody PBP1510 in Patients With Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prestige Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PAUF-I; 2024-514379-16-00 (EU CTIS Number); 2021-000682-32 (EudraCT Number)
Record Dates: First submitted 2021-08-27; First posted 2021-12-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Cohort 1M (Experimental): 1 mg/kg of PBP1510 as monotherapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL)
- Cohort 1C (Experimental): 1 mg/kg of PBP1510 and 1000 mg/m^2 of gemcitabine as combination therapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL); Drug: Gemcitabine (1000 mg/m^2)
- Cohort 2M (Experimental): 3 mg/kg of PBP1510 as monotherapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL)
- Cohort 2C (Experimental): 3 mg/kg of PBP1510 and 1000 mg/m^2 of gemcitabine as combination therapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL); Drug: Gemcitabine (1000 mg/m^2)
- Cohort 3M (Experimental): 6 mg/kg of PBP1510 as monotherapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL)
- Cohort 3C (Experimental): 6 mg/kg of PBP1510 and 1000 mg/m^2 of gemcitabine as combination therapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL); Drug: Gemcitabine (1000 mg/m^2)
- Cohort 4M (Experimental): 10 mg/kg of PBP1510 as monotherapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL)
- Cohort 4C (Experimental): 10 mg/kg of PBP1510 and 1000 mg/m^2 of gemcitabine as combination therapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL); Drug: Gemcitabine (1000 mg/m^2)
- Cohort 5M (Experimental): 15 mg/kg of PBP1510 as monotherapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL)
- Cohort 5C (Experimental): 15 mg/kg of PBP1510 and 1000 mg/m^2 of gemcitabine as combination therapy will be administered
  Interventions: Drug: PBP1510 (400mg/16mL); Drug: Gemcitabine (1000 mg/m^2)

INTERVENTIONS:
Drug: PBP1510 (400mg/16mL) — Humanized immunoglobulin G1 (IgG1) monoclonal antibody (mAb) that targets and neutralizes PAUF, administered as a 90-minute intravenous infusion
Drug: Gemcitabine (1000 mg/m^2) — Humanized immunoglobulin G1 (IgG1) monoclonal antibody (mAb) that targets and neutralizes PAUF, administered as a 90-minute intravenous infusion in combination with 1000 mg/m2 gemcitabine administered as a 30-minute intravenous infusion.
  Arms: Cohort 1C; Cohort 2C; Cohort 3C; Cohort 4C; Cohort 5C

SUMMARY:
The first in human clinical study is planned as an open-label, dose-escalation, and dose-expansion, multicentre, two-part, Phase 1/2a study of PBP1510 administered to patients with advanced/metastatic pancreatic cancer. The study will be conducted in two parts, Part 1 as a PBP1510 single agent dose-escalation, and PBP1510 dose-escalation in combination with gemcitabine, and Part 2 as PBP1510 dose-expansion at the RP2D in combination with gemcitabine.

DETAILED DESCRIPTION:
The first in human clinical study is planned as an open-label, multicentre, two-part, Phase 1/2a study to assess the safety, pharmacokinetics, and efficacy of PBP1510 in patients with advanced/metastatic pancreatic cancer. Part 1 (Phase 1) is a dose-escalation phase, wherein PBP1510 will be administered, as monotherapy (monotherapy cohorts) or in combination with gemcitabine (combination cohorts) in advanced/metastatic pancreatic cancer patients whose tumours have progressed on at least one previous line of chemotherapy for locally advanced/metastatic disease. The RP2D will be selected based on the analysis of the PK, safety, and efficacy data. Part 2 (Phase 2a) will be an open-label study and patients will be administered the RP2D of PBP1510 derived from Part 1, in combination with gemcitabine for advanced/metastatic pancreatic cancer patients whose tumour has progressed on one previous line of chemotherapy for locally advanced/metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolling into Part 1 (Phase 1), or Part 2 (Phase 2a) must meet all of the following inclusion criteria:

1. Adults ≥ 18 years of age (or the legal age of majority in the country of recruitment) at the time consent is obtained.
2. Patient should understand, voluntarily sign, and date the written consent form prior to any protocol-specific procedures.
3. Performance Status score less than or equal to 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
4. Have histological or cytological evidence of a diagnosis of pancreatic cancer that is advanced and/or metastatic.
5. Have a life expectancy of ≥ 3 months.
6. No other malignancy present that would interfere with the current intervention.
7. Prior radiation therapy for treatment of cancer is allowed to < 25% of the bone marrow, and patients must have recovered from the acute toxic effects of their treatment prior to study enrolment. Prior radiotherapy must be completed at least 4 weeks before the first dose of study treatment.
8. At least one measurable lesion as per RECIST v1.1
9. Adequate baseline organ function defined as:

   ANC ≥ 1.5 × 10^9 /L; Haemoglobin ≥ 9 g/dL; Platelets ≥ 100 × 10^9 /L; Total bilirubin ≤ 2 × ULN (≤ 3 x ULN for patients with biliary stenting and patients with Gilbert's syndrome); AST and ALT < 3 x ULN (≤ 5 x ULN for patients with hepatic metastases); Serum creatinine OR creatinine clearance (as determined by the Cockcroft Gault formula) OR eGFR based on MDRD ≤ 1.5 x ULN OR ≥ 50 mL/min OR ≥ 50 mL/min/1.73 m^2; LVEF ≥ 50% by ECHO or MUGA; QTc ≤ 470 ms
10. Female patients of nonchildbearing potential must meet at least 1 of the following criteria: have undergone a documented hysterectomy, and/or bilateral oophorectomy; have medically confirmed ovarian failure or achieved postmenopausal status. A postmenopausal state is defined as cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause and have a follicle stimulating hormone (FSH) level confirming the postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. Female patients of childbearing potential must have a negative serum pregnancy test within 28 days prior to and negative urine pregnancy test just prior to the first dose of PBP1510 and agree to use effective contraception, in accordance with the recommendations of the Clinical Trials Facilitation and Coordination Group (CTFG) from study entry and until for at least 6 months after the last dose of PBP1510.
11. For women of childbearing potential and men with partners of childbearing potential, agreement (by patient and/or partner) to use two effective forms of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) from study entry and until for at least 6 months after the last dose of PBP1510.

    Investigator or his/her representative should discuss acceptable pregnancy prevention method(s) with the patients. Highly effective methods of birth control include those that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, levonorgestrel-releasing intrauterine system, intra-uterine devices (IUDs), and true sexual abstinence.
12. Patients must be willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.

    Patients enrolling into Part 1 (Phase 1) of the study must also meet the following inclusion criteria:
13. Monotherapy and combination cohorts: advanced/metastatic pancreatic cancer patients whose tumours have progressed after at least one prior line of standard chemotherapy.

    Patients enrolling into Part 2 (Phase 2a) of the study must also meet the following inclusion criteria:
14. Advanced/metastatic pancreatic cancer patients whose tumours have progressed after one prior line of standard chemotherapy.

Exclusion Criteria:

Patients enrolling into Part 1 (Phase 1), or Part 2 (Phase 2a) will be excluded if any of the following criteria apply:

1. Patients who have known brain metastases will be excluded from the study. However, a patient may be included in the study, if has been previously treated for brain metastasis, the disease is well controlled for at least 3 months, and the patient is off steroids.
2. Patients who have undergone a major surgery within 4 weeks prior to the start of PBP1510 administration, other than endoscopic/radiation procedures, bypass surgery (i.e., gastrojejunostomy), laparoscopy, port placement or a diagnostic surgery (i.e., surgery done to obtain a diagnostic biopsy, without removal of an organ), as long as the patient has recovered from these minor surgical procedures.
3. Patients who have active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, e.g., an active opportunistic infection with mycobacteria, cytomegalovirus, toxoplasma, Pneumocystis carinii (P. carinii), or other microorganisms that is under treatment with myelotoxic drugs.
4. Patient has a known history of human immunodeficiency virus (HIV; HIV 1/2 antibodies).
5. Patient has known history of or currently active hepatitis B (e.g., hepatitis B antigen [HBsAg] reactive), hepatitis C (e.g., HCV RNA [qualitative] is detected) or syphilis [Venereal Disease Research Laboratory (VDRL) to detect antibodies in blood]).
6. Patient has impaired cardiac function and uncontrolled cardiac diseases/hypertension that are deemed clinically significant by the Investigator and which could compromise the patient's safety or the study data integrity.
7. Patient has serious psychiatric disorders, which could compromise the patient's safety or the study data integrity.
8. Any other malignancy from which the patient has been disease-free for less than 5 years, except for adequately treated and cured basal or squamous cell skin cancer.
9. Patients who are enrolled in any other therapeutic clinical trial.
10. Patients currently receiving radiation therapy or those having received radiation within 4 weeks prior to study entry.
11. Patients having received investigational anti-cancer drug within 28 days (or 5 half-lives, whichever is longer) preceding the first dose of PBP1510 or chemotherapy within the last 4 weeks prior to the first dose of PBP1510.
12. Patients with known allergy or hypersensitivity to components of the PBP1510 formulation including the excipients and history of hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
13. Patients who are pregnant, or breast feeding.
14. Patients who are unwilling or unable to comply with study procedures.
15. Patients who are not eligible to participate in this study, as judged by Investigators.
16. A history of allergic reactions attributed to gemcitabine or compounds of similar chemical composition to gemcitabine and/or previous treatment discontinuation due to gemcitabine toxicity.

Note: Patients with previous exposure to gemcitabine should not be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PART 1 (PHASE 1): To evaluate safety and tolerability of PBP1510 | Baseline to Safety Follow Up visit (90 days after last dose of PBP1510)
  As assessed by evaluation of adverse events and serious adverse events (AE & SAE). AEs will be coded using MedDRA and grouped by system organ class and preferred term. An AE which is fatal or life threatening will be considered as SAE.
PART 1 (PHASE 1): Dose limiting toxicity (DLT) evaluation | During first treatment cycle (each cycle is 28 days)
  DLTs will be assessed by the Investigator using the NCI-CTCAE V5.0.
PART 2 (PHASE 2a): To establish safety of PBP1510 in combination with gemcitabine | Baseline to Safety Follow Up visit (90 days after last dose of PBP1510)
  As assessed by evaluation of AEs and SAEs. AEs will be coded using MedDRA and grouped by system organ class and preferred term. An AE which is fatal or life threatening will be considered as SAE.
PART 2 (PHASE 2a): To assess the efficacy of PBP1510 in combination with gemcitabine | Baseline to End of Treatment visit (28 days after last dose of PBP1510)
  As assessed by objective response rate (ORR; rate of patients with complete response [CR] or partial response [PR]) evaluated by Response Evaluation Criteria in Solid Tumours version v1.1 (RECIST v1.1).
PART 1 (PHASE 1): Determine the recommended Phase 2a dose (R2PD) of PBP1510 | After last patient enrolled in last dosing cohort completes 4 cycles of treatment. Each cycle is 28 days.
  The RP2D will be selected based on the analysis of the PK, safety, and efficacy data.

SECONDARY OUTCOMES:
PART 1 (PHASE 1): Peak concentration (Cmax) of PBP1510 (µg/ml) | Cycle (C) 1 Day (D) 1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Time to reach Cmax (Tmax) of PBP1510 (hr) | C1D1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Terminal elimination half-life (t1/2) of PBP1510 (hr) | C1D1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Area under the concentration-time curve (AUC) of PBP1510 (hr*µg /ml) | C1D1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Mean residence time (MRT) of PBP1510 (hr) | C1D1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Volume of distribution at steady state (Vss) of PBP1510 (mL/kg) | C1D1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Volume of the central compartment (Vc) of PBP1510 (mL/kg) | C1D1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Clearance (CL) of PBP1510 (mL/kg/hr) | C1D1, C1D2, C1D3, C1D5, C1D8, C1D15, C1D22, C2D1, C2D8, C2D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered as monotherapy, and in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease
PART 1 (PHASE 1): Peak concentration (Cmax) of gemcitabine (µg/ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 1 (PHASE 1): Time to reach Cmax (Tmax) of gemcitabine (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 1 (PHASE 1): Terminal elimination half-life (t1/2) of gemcitabine (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 1 (PHASE 1): Area under the concentration-time curve (AUC) of gemcitabine (hr*µg /ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 1 (PHASE 1): Mean residence time (MRT) of gemcitabine (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 1 (PHASE 1): Clearance (CL) of gemcitabine (mL/kg/hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 1 (PHASE 1): Presence of anti-drug antibody (ADA) and neutralizing antibodies (NAb) against PBP1510 administered as monotherapy, and in combination with gemcitabine. | C1D1, C1D15, C2D1, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Trough concentration (Ctrough) of PBP1510 (µg/ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Peak concentration (Cmax) of PBP1510 (µg/ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Time to reach Cmax (Tmax) of PBP1510 (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Terminal elimination half-life (t1/2) of PBP1510 (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Area under the concentration-time curve (AUC) of PBP1510 (hr*µg /ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Mean residence time (MRT) of PBP1510 (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Volume of distribution at steady state (Vss) of PBP1510 (mL/kg) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Volume of the central compartment (Vc) of PBP1510 (mL/kg) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Clearance (CL) of PBP1510 (mL/kg/hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow Up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  administered in combination with gemcitabine, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Trough concentration (Ctrough) of Gemcitabine (µg/ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Peak concentration (Cmax) of Gemcitabine (µg/ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Time to reach Cmax (Tmax) of Gemcitabine (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Terminal elimination half-life (t1/2) of Gemcitabine (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Area under the concentration-time curve (AUC) of Gemcitabine (hr*µg /ml) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Mean residence time (MRT) of Gemcitabine (hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Clearance (CL) of Gemcitabine (mL/kg/hr) | C1D1, C1D8, C1D15, C2D1, C2D8, C2D15, C3D1, C3D8, C3D15, C4D1, C4D8, C4D15. Each cycle is 28 days.
  administered in combination with PBP1510, following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Progression-free survival (PFS) after treatment with PBP1510 administered in combination with gemcitabine | From the first PBP1510 infusion to date of first documentation of progressive disease or death from any cause, through study completion (approximately 1 year)
  in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Overall Survival (OS) after treatment with PBP1510 administered in combination with gemcitabine | From the first PBP1510 infusion to the date of death due to any cause, through study completion (approximately 1 year)
  in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Duration of Response (DoR) after treatment with PBP1510 administered in combination with gemcitabine | from the first documentation of overall response (CR or PR) post first PBP1510 infusion to the first documentation of disease progression or death from any cause, through study completion (approximately 1 year)
  in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a): Presence of ADA and NAb against PBP1510 administered in combination with gemcitabine. | C1D1, C2D1, C3D1, C4D1, End of Treatment visit (28 days after last dose of PBP1510) and Safety Follow-up visit (90 days after last dose of PBP1510). Each cycle is 28 days.
  following IV administration, in patients with pancreatic cancer whose tumours have progressed after one previous line of chemotherapy for locally advanced/metastatic disease.

OTHER OUTCOMES:
PART 1 (PHASE 1) Exploratory Endpoint: Preliminary evidence of clinical outcomes as assessed by objective response rate (ORR) after treatment with PBP1510 administered as monotherapy, and in combination with gemcitabine. | Through study completion (approximately 1 year)
  following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 1 (PHASE 1) Exploratory Endpoint: Analysis of PAUF in tumour tissue pre-treatment and after treatment with PBP1510 administered as monotherapy, and in combination with gemcitabine. | Through study completion (approximately 1 year)
  following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a) Exploratory Endpoint: Pre-treatment PAUF expression and clinical efficacy outcome after treatment with PBP1510 administered in combination with gemcitabine. | Through study completion (approximately 1 year)
  following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.
PART 2 (PHASE 2a) Exploratory Endpoint: Analysis of PAUF in tumour tissue pre-treatment and after treatment with PBP1510 administered in combination with gemcitabine. | Through study completion (approximately 1 year)
  following IV administration, in patients with pancreatic cancer whose tumours have progressed after at least one previous line of chemotherapy for locally advanced/metastatic disease.

CONTACTS AND LOCATIONS:
Locations (4):
- Northwell Health / R.J. Zuckerberg Cancer Center, New Hyde Park, New York, United States
- Monash Health, Melbourne, Australia
- National Cancer Centre Singapore, Singapore, Singapore
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No